CLINICAL TRIAL: NCT04685525
Title: Mycobiome Supporting Diet (MSD) to Reduce Gastrointestinal (GI) Toxicity Associated With Autologous Stem Cell Transplant (ASCT) For Patients With Multiple Myeloma (MM)
Brief Title: Mycobiome Supporting Diet to Reduce GI Toxicity Associated With ASCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative decision
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE12Z20
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Autologous Transplant; Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mycobiome Supporting Diet (Experimental): Participants will be able to abide by the allowed and disallowed foods in MSD diet for at least four consecutive weeks prior to conditioning and up to 10 days after transplant. Participants will maintain a diary of foods they consume and any adverse effects they are experiencing and will self- collect fecal samples 28 days before transplant, 2 days before transplant and 10 days after transplant
  Interventions: Behavioral: Mycobiome Supporting Diet

INTERVENTIONS:
Behavioral: Mycobiome Supporting Diet — MSD takes combines elements from several diets (e.g., Paleo, low-carbohydrate, vegetarian, and Mediterranean) and excludes elements of these diets that have been specifically proven to increase pathogenic fungi in the human gut.

SUMMARY:
The purpose of this study is to determine if this specific Mycobiome Supporting Diet (MSD diet) can help reduce gut inflammation during post-transplant period. The MSD is an special diet which will be explained in detail by a dietician that works by supporting the body's good gut bacteria and fungi.

DETAILED DESCRIPTION:
This is a non-randomized cohort study. Participants will be on a specific diet for 4 weeks prior to transplant and 10 days after transplant, and will then be asked to fill out several questionnaires during this period to see if this diet is easy and simple to follow. The questionnaires will be weekly while participants are outpatient and once admitted to the hospital, participants will need to fill it on the last day (10 days after stem cell infusion). Participants will also be requested to provide fecal swab samples which we will test for bacteria and fungi. A total of 3 samples will be taken at different time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for first autologous transplant for myeloma
* Willing to adhere to the allowed and disallowed foods of the diet plan.
* Able to get and prepare their own food items for all meals during the study

Exclusion Criteria:

* Active inflammatory bowel disease, celiac disease, other chronic intestinal disorders
* Pregnant women, planning to get pregnant or breastfeeding
* Prior bowel resection
* Inability to tolerate the study diet due to allergies/ intolerance/ preference
* Inability to consent to trial
* Patients with restrictions in diet including inability to have oral nutrition with regular consistency
* Any condition that the investigator feels may limit the volunteer's ability to complete the study protocol.
* Patients with absolute neutrophil count (ANC) < 1000 on long term antibacterial prophylaxis ongoing 3 days prior to enrollment
* Patients who received antifungal therapy in 3 days prior to enrollment
* Patients who received steroid therapy in 7 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire | 21 days prior to Transplant (an average of 1 month from start of study)
  MSD adherence feasibility measured by percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire. The questionnaire includes a multiple choice questions about adherence to diet (4 levels, from 'not at all' to 'the whole time'), a multiple choice question identifying barriers to adherence, and 8 yes/no questions about medication use and symptom experience. The MSD diet will deem feasible if at least 80 percent of participants showed adherence defined by 2 out of 3 assessment marked "more than half the time".
Percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire | 14 days prior to transplant (an average of 1 month from start of study)
  MSD adherence feasibility measured by percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire. The questionnaire includes a multiple choice questions about adherence to diet (4 levels, from 'not at all' to 'the whole time'), a multiple choice question identifying barriers to adherence, and 8 yes/no questions about medication use and symptom experience. The MSD diet will deem feasible if at least 80 percent of participants showed adherence defined by 2 out of 3 assessment marked "more than half the time".
Percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire | 7 days prior to transplant (an average of 1 month from start of study)
  MSD adherence feasibility measured by percent of participants with at least 2 out of 3 assessments marked "more than half the time" on compliance questionnaire. The questionnaire includes a multiple choice questions about adherence to diet (4 levels, from 'not at all' to 'the whole time'), a multiple choice question identifying barriers to adherence, and 8 yes/no questions about medication use and symptom experience. The MSD diet will deem feasible if at least 80 percent of participants showed adherence defined by 2 out of 3 assessment marked "more than half the time".
Patient-reported outcome (PRO)-Common Terminology Criteria for Adverse Even CTCAE questionnaire | After baseline (7 days post-transplant)
  Patient perception of symptoms measured using PRO-CTCAE questionnaire, consisting of 15 questions with frequency and severity scores, questions ranging 1 to 5, 5 is worse and 1 is less
PRO-CTCAE questionnaire scores | week 1 in the 1 month prior to transplant
  Patient perception of symptoms measured using PRO-CTCAE questionnaire, consisting of 15 questions with frequency and severity scores, questions ranging 1 to 5, 5 is worse and 1 is less
PRO-CTCAE questionnaire scores | week 2 in the 1 month prior to transplant
  Patient perception of symptoms measured using PRO-CTCAE questionnaire, consisting of 15 questions with frequency and severity scores, questions ranging 1 to 5, 5 is worse and 1 is less
PRO-CTCAE questionnaire scores | week 3 in the 1 month prior to transplant
  Patient perception of symptoms measured using PRO-CTCAE questionnaire, consisting of 15 questions with frequency and severity scores, questions ranging 1 to 5, 5 is worse and 1 is less
PRO-CTCAE questionnaire scores | week 4 in the 1 month prior to transplant
  Patient perception of symptoms measured using PRO-CTCAE questionnaire, consisting of 15 questions with frequency and severity scores, questions ranging 1 to 5, 5 is worse and 1 is less

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Malek, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the small sample size of the study participants in order to protect their identities.